CLINICAL TRIAL: NCT01974284
Title: Percutaneous Ethanol Injection for Primary Papillary Thyroid Microcarcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient enrollment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIC1312013168
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Administration, Cutaneous; Ethanol; Thyroid (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- percutaneous ethanol ablation (Experimental): The experimental group of the study is comprised of patients that will undergo percutaneous ethanol ablation for the management of papillary thyroid microcarcinoma.
  Interventions: Drug: percutaneous ethanol ablation

INTERVENTIONS:
Drug: percutaneous ethanol ablation — The volume of 99% ethanol to be injected is calculated using a standardized formula. Ethanol is instilled with a needle under ultrasound guidance after administration of local anesthesia.
  Other Names: percutaneous; ethanol; ablation; papillary; thyroid; microcarcinoma; PTMC

SUMMARY:
We assess the effectiveness of percutaneous ethanol ablation for the treatment of thyroid cancer.

DETAILED DESCRIPTION:
We hypothesize that percutaneous ethanol ablation (PEA) for primary papillary thyroid microcarcinoma (PTMC) has equivalent oncologic outcomes to current treatment options including observation, thyroid lobectomy and total thyroidectomy. In addition, we hypothesize that it will yield superior long-term quality of life, including measures of pain, voice, and cosmesis than standard surgical therapy (total thyroidectomy). If our hypotheses are correct, the findings of this study have the potential to fundamentally change clinical management of this group of patients.

This study was changed from its initial design: a 2 arm study comparing PEA to surgery (Amended April 30, 2015). The change in design was made based on several discussions within Yale Endocrine Surgery, with patients diagnosed with PTMC, and knowledge of other institutions performing PEA for PTMC as standard of care.

The study team had been contacted by numerous potential subjects interested in PEA who were unwilling to be randomized to surgery. Because patients interested in PEA appeared to be firmly against the idea of thyroidectomy, we believed that we would be unable to enroll sufficient patients to this study as the protocol originally stood.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis: single, cytology-proven papillary thyroid carcinoma measuring 1 cm or less in diameter (microcarcinoma, T1a), without visible extrathyroidal extension, and with negative central and lateral neck lymph nodes by ultrasound

Exclusion Criteria:

* Patient refusal to participate
* History of prior thyroid or parathyroid surgery
* Previous recurrent laryngeal nerve injury
* Inability to make decisions or comply with follow up
* Co-existing indication for thyroidectomy
* Aggressive cytological or molecular features
* Multifocal papillary thyroid carcinoma
* Pregnant or breast-feeding
* Anatomically unfavorable location of the tumor (proximity to recurrent laryngeal nerve or trachea)
* Documented or suspected distant metastasis
* History of radiation to neck or face
* Family history of thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03-02 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Callender, MD, Principal Investigator — Yale University- Department of Surgery
Locations (1):
- Endocrine Surgery Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Percutaneous Ethanol Ablation
Started | 7
Completed | 0
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: 7 patients enrolled in the study.
Arm/Group | Percutaneous Ethanol Ablation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Disease-free
Description: Primary endpoint of the study consists of the oncological outcome, which includes the disease-free status of the patients.
Time Frame: 5 years
Population: Patients were not followed as the study was terminated.
Arm/Group | Percutaneous Ethanol Ablation
Number analyzed (Participants) | 0

2. Primary Outcome: Overall Survival
Description: Primary endpoint of the study consists of the oncological outcome, which includes the overall survival of the patients.
Time Frame: 5 years
Population: Patients were not followed as the study was terminated.
Arm/Group | Percutaneous Ethanol Ablation
Number analyzed (Participants) | 0

3. Secondary Outcome: Quality of Life
Description: The Short-Form-36 (SF-36) health survey is a patient-reported survery that evaluates the patient's health status. It consists of 8 scaled scores which are the weighted sums of the questions in each section. The 8 sections that are tested are vitality, physical functioning, bodily pain, general role functioning, emotional role functioning, social role functioning, and mental health. Each scale is directly transformed into a 0-100 scale; the higher the score, the less disability (i.e. the score of 0 is equivalent to maximal disability, and the score of 100 is equivalent of no disability). The SF-36 is a set of easily-administered quality-of-life measures and is a validated tool to evaluate patient quality of life.
Time Frame: 5 years
Population: Patients were not followed as the study was terminated.
Arm/Group | Percutaneous Ethanol Ablation
Number analyzed (Participants) | 0

4. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction will be assessed by evaluating the following: pain with the "Brief Pain Inventory" (BPI), voice with the "Voice Handicap Index" (VHI) and cosmesis with the "Patient and Observer Scar Assessment Scale" (POSAS). The BPI is a simple, well-accepted instrument for the objective assessment of pain. The VHI is an established tool used to assess voice after an intervention. POSAS is a validated tool for the evaluation of surgical scars.
Time Frame: 5 years
Population: Patients were not followed as the study was terminated.
Arm/Group | Percutaneous Ethanol Ablation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored until the time of study termination.
Arm/Group | Percutaneous Ethanol Ablation
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT01974284/Prot_SAP_000.pdf